CLINICAL TRIAL: NCT00029900
Title: Phase I Testing of ADI-PEG in Metastatic Melanoma
Brief Title: ADI-PEG in Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: FDA Office of Orphan Products Development (U.S. Federal Agency)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: FD-R-2003-01; FD-R-002003-01
Record Dates: First submitted 2002-01-24; First posted 2002-01-25 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2002-01

CONDITIONS: Melanoma; Neoplasm Metastasis
Keywords: Dose-Response Relationship, Drug; Polyethylene Glycol; Arginine Deiminase
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis | interventions — ADI PEG20

INTERVENTIONS:
Drug: ADI PEG

SUMMARY:
This is a study to determine the safety and toxicity of increasing doses of arginine deiminase combined to polyethylene glycol (ADI-PEG) in patients with nonresectable metastatic melanoma.

DETAILED DESCRIPTION:
The use of amino acid degrading enzymes derived from microbial sources has proven to be an effective means of controlling some forms of cancer auxotrophic for nonessential amino acids. Recently it has been shown that human melanomas are auxotrophic for arginine. As arginine is a nonessential amino acid for humans, elimination of it may prove to be an effective method for controlling cancer. Laboratory studies have provided promising results with the arginine-degrading enzyme arginine deiminase (ADI) coupled to polyethylene glycol (PEG) to enhance its circulating half-life.

In this study, patients each receive 3 intramuscular treatments of ADI-SS PEG over a 4-week period. There are 4 cohorts of patients each receiving a different dose level. Pharmacokinetics, pharmacodynamics, safety and toxicity, and immunogenicity studies will be performed.

ELIGIBILITY:
Inclusion criteria:

* Histologically confirmed metastatic melanoma
* Nonresectable disease
* Measurable or evaluable disease
* Progressive disease following standard chemotherapy, radiotherapy, surgery, or immunotherapy; and no longer responding to therapy
* Recovered from prior surgery
* Karnofsky performance status 70 or higher
* Expected survival of at least 12 weeks
* Bilirubin less than 2.0 mg/dL
* Albumin greater than 3.0 g/dL
* SGOT less than 5 times upper limit of normal (ULN)
* Alkaline phosphatase less than 5 times ULN
* Ammonia less than 55 microg/dL
* Glucose greater than 60 mg/dL
* Amylase less than 1.5 times ULN
* Absolute neutrophil count greater than 1,500/mm3
* Platelet count greater than 100,000/mm3
* Patients must use 2 forms of effective contraception

Exclusion criteria:

* Prior therapy within the past 4 weeks
* Ascites or pleural effusion
* Significant cardiac disease (i.e., New York Heart Association class III or IV heart disease)
* Pregnant or nursing
* Concurrent enrollment in another IND study
* Serious infection requiring antibiotics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15
Dates: Start 2001-09; Study Completion 2003-08

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States